CLINICAL TRIAL: NCT04179474
Title: A Phase 1b, Two-Part, Open-Label, Fixed-Sequence, Safety, Tolerability and Drug-Drug Interaction Study Between Single Dose Erenumab or Galcanezumab and Multiple Dose Ubrogepant in Participants With Migraine
Brief Title: Safety, Tolerability and Drug- Drug Interaction Study of Ubrogepant With Erenumab or Galcanezumab in Participants With Migraine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 3110-108-002
Record Dates: First submitted 2019-09-26; First posted 2019-11-27 (Actual); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Migraine
Keywords: ubrogepant; erenumab; galcanezumab; safety; tolerability; interaction
MeSH Terms: conditions — Migraine Disorders | interventions — ubrogepant; erenumab; galcanezumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Intervention A then B then D) (Experimental): Intervention A: Single oral dose of ubrogepant 100 mg tablet on Day 1 under fasted conditions; followed by Intervention B: Single subcutaneous (SC) injection of erenumab 140 mg on Day 8; followed by Intervention D: Ubrogepant 100 mg tablet orally once daily on Days 12, 13, 14 and 15 under fasted conditions.
  Interventions: Drug: Ubrogepant; Drug: Erenumab
- Part 2 (Intervention A then C then D) (Experimental): Intervention A: Single oral dose of ubrogepant 100 mg tablet on Day 1 under fasted conditions; followed by Intervention C: Two SC injections of galcanezumab 120 mg on Day 8; followed by Intervention D: Ubrogepant 100 mg tablet orally once daily on Days 12, 13, 14 and 15 under fasted conditions.
  Interventions: Drug: Ubrogepant; Drug: Galcanezumab

INTERVENTIONS:
Drug: Ubrogepant — Oral administration of 100 mg ubrogepant tablet once daily [Intervention A=single dose and Intervention D=repeated daily dose].
Drug: Erenumab — Single dose subcutaneous (SC) injection of erenumab 140 mg [Intervention B].
  Arms: Part 1 (Intervention A then B then D)
Drug: Galcanezumab — 2 SC injections of galcanezumab 120 mg [Intervention C].
  Arms: Part 2 (Intervention A then C then D)

SUMMARY:
This study will evaluate the potential for a pharmacokinetic (PK) interaction and provide safety and tolerability information when ubrogepant and erenumab or ubrogepant and galcanezumab are co-administered.

ELIGIBILITY:
Inclusion Criteria:

* At least a 1-year history of migraine with or without aura consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd edition, (ICHD-3, 2018)
* By history, the participant's migraines typically last between 4 and 72 hours if untreated or treated unsuccessfully and migraine episodes are separated by at least 48 hours of headache pain freedom
* History of at least 2 migraine attacks per month in the 2 months prior to Screening
* Have a sitting pulse rate ≥ 45 beats per minute (bpm) and ≤ 100 bpm during the vital sign assessment at the Screening Visit. Clinical site may perform a maximum of 2 repeats of vital sign measurements if the initial measurement is out of range.
* Negative test results for benzoylecgonine (cocaine), methadone, barbiturates, amphetamines, benzodiazepines, cannabinoids, opiates, and phencyclidine at the Screening Visit and Day -1; unless explained by concomitant medication use (eg, opioids prescribed for migraine pain)
* Participants willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period

Exclusion Criteria:

* Difficulty distinguishing migraine headache from tension-type or other headaches
* Has a history of migraine aura with diplopia or impairment of level of consciousness, hemiplegic migraine, or retinal migraine as defined by ICHD-3
* Has a current diagnosis of new persistent daily headache, trigeminal autonomic cephalgia (eg, cluster headache), or painful cranial neuropathy as defined by ICHD-3
* Required hospital treatment of a migraine attack 3 or more times in the 6 months prior to Screening
* Has a chronic non-headache pain condition requiring daily pain medication (with the exception of pregabalin)
* Has clinically significant cardiovascular or cerebrovascular disease per the investigator's opinion
* Previously participated in an investigational study of ubrogepant
* Participation in any other clinical investigation using an experimental drug within 30 days prior to study intervention administration
* Participation in a blood or plasma donation program within 60 or 30 days, respectively, prior to study intervention administration

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Boinpally, Study Director — Allergan
Locations (2):
- United States (2):
  - QPS, Springfield, Missouri
  - Spaulding, West Bend, Wisconsin

REFERENCES:
- [Result] Jakate A,Boinpally R, Butler M, Borbridge L, Contreras-De Lama J, McGeeney D, Periclou A. Safety and tolerability of ubrogepant for the acute treatment of migraine following co-administration with preventive monoclonal antibody treatment [abstract]. In:62nd Annual Scientific Meeting American Headache Society; June2020; San Diego, California.

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1 (First Intervention)
Arm/Group | Part 1 (Intervention A Then B Then D) | Part 2 (Intervention A Then C Then D)
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Treatment Period 2 (Second Intervention)
Arm/Group | Part 1 (Intervention A Then B Then D) | Part 2 (Intervention A Then C Then D)
Started | 19 (1 participant did not receive Intervention B.) | 20
Completed | 19 | 20
Not Completed | 0 | 0
Period: Treatment Period 3 (Third Intervention)
Arm/Group | Part 1 (Intervention A Then B Then D) | Part 2 (Intervention A Then C Then D)
Started | 19 | 19 (1 participant did not receive Intervention D.)
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received/took at least 1 administration of study intervention in Part 1 or Part 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 (Intervention A Then B Then D) | Part 2 (Intervention A Then C Then D) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Customized [Mean (Full Range); unit: years] | 32.2 [20 to 50] | 38.4 [18 to 50] | 35.3 [18 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 10 | 8 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 20 | 16 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 12 | 11 | 23
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Plasma Concentration Versus Time Curve From Time 0 to Time t (AUC0-t) for Ubrogepant Alone and in Combination With Erenumab
Time Frame: Day 1 (Treatment Period 1): Predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 14, and 24 hours postdose; Day 12 (Day 1 of Treatment Period 3): Predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 14, and 24 hours postdose
Population: Pharmacokinetic 1 (PK1) population included all participants who had evaluable plasma PK parameters of ubrogepant for both ubrogepant alone and ubrogepant in combination with erenumab or galcanezumab.
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*h/mL)
Groups:
- Part 1: Ubrogepant Alone: Participants received Intervention A (ubrogepant 100 mg tablet) single oral dose on Day 1 under fasted conditions.
- Part 1: Ubrogepant in Combination With Erenumab: Participants received Intervention B: SC injection of erenumab 140 mg on Day 8; followed by Intervention D: Ubrogepant 100 mg tablet orally on Day 12 under fasted conditions.
Arm/Group | Part 1: Ubrogepant Alone | Part 1: Ubrogepant in Combination With Erenumab
Number analyzed (Participants) | 20 | 19
nanogram*hour/milliliter (ng*h/mL) | 1841.42 (490.17) | 1959.96 (639.51)
Statistical Analysis 1: Comparison: Part 1: Ubrogepant Alone vs Part 1: Ubrogepant in Combination With Erenumab; A linear mixed-effects model with study intervention as fixed effect and participant as a random effect was used to determine the Geometric Means; Test type: Equivalence — "No effect" of co-administration with erenumab on the PK of ubrogepant was concluded if the 90% CIs for the geometric mean ratios of ubrogepant PK parameters for test study intervention (ubrogepant in combination with erenumab) versus reference study intervention (ubrogepant alone) were within the limits of 80% to 125%; Ratio of Geometric Mean Percentage = 105.55, 90% CI 2-sided [96.21 to 115.79] — Ratio of Geometric Mean Percentage=Ubrogepant in Combination with Erenumab/Ubrogepant Alone * 100

2. Primary Outcome: Part 2: AUC0-t for Ubrogepant Alone and in Combination With Galcanezumab
Time Frame: as for outcome 1
Population: PK1 population included all participants who had evaluable plasma PK parameters of ubrogepant for both ubrogepant alone and ubrogepant in combination with erenumab or galcanezumab
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Part 2: Ubrogepant Alone: Participants received Intervention A (ubrogepant 100 mg tablet) orally once daily on Day 1 under fasted conditions.
- Part 2: Ubrogepant in Combination With Galcanezumab: Participants received Intervention C: Two SC injections of galcanezumab 120 mg on Day 8; followed by Intervention D: Ubrogepant 100 mg tablet orally on Day 12 under fasted conditions.
Arm/Group | Part 2: Ubrogepant Alone | Part 2: Ubrogepant in Combination With Galcanezumab
Number analyzed (Participants) | 20 | 19
ng*h/mL | 1700.31 (913.42) | 1758.05 (1033.44)
Statistical Analysis 1: Comparison: Part 2: Ubrogepant Alone vs Part 2: Ubrogepant in Combination With Galcanezumab; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — "No effect" of co-administration with galcanezumab on the PK of ubrogepant was concluded if the 90% CIs for the geometric mean ratios of ubrogepant PK parameters for test study intervention (ubrogepant in combination with galcanezumab) versus reference study intervention (ubrogepant alone) were within the limits of 80% to 125%; Ratio of Geometric Mean Percentage = 105.03, 90% CI 2-sided [89.55 to 123.19] — Ratio of Geometric Mean Percentage=Ubrogepant in Combination with Galcanezumab/Ubrogepant Alone * 100

3. Primary Outcome: Part 1: Area Under the Plasma Concentration Versus Time Curve From Time 0 to Infinity (AUC0-∞) for Ubrogepant Alone and in Combination With Erenumab
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Part 1: Ubrogepant Alone | Part 1: Ubrogepant in Combination With Erenumab
Number analyzed (Participants) | 20 | 19
ng*h/mL | 1878.25 (497.82) | 1993.40 (639.22)
Statistical Analysis 1: Comparison: Part 1: Ubrogepant Alone vs Part 1: Ubrogepant in Combination With Erenumab; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Mean Percentage = 105.38, 90% CI 2-sided [96.19 to 115.45] — Ratio of Geometric Mean Percentage=Ubrogepant in Combination with Erenumab/Ubrogepant Alone * 100

4. Primary Outcome: Part 2: AUC0-∞ for Ubrogepant Alone and in Combination With Galcanezumab
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Part 2: Ubrogepant Alone | Part 2: Ubrogepant in Combination With Galcanezumab
Number analyzed (Participants) | 20 | 19
ng*h/mL | 1732.22 (928.06) | 1793.74 (1057.02)
Statistical Analysis 1: Comparison: Part 2: Ubrogepant Alone vs Part 2: Ubrogepant in Combination With Galcanezumab; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of Geometric Mean Percentage = 104.76, 90% CI 2-sided [89.68 to 122.38] — Ratio of Geometric Mean Percentage=Ubrogepant in Combination with Galcanezumab/Ubrogepant Alone * 100

5. Primary Outcome: Part 1: Maximum Plasma Drug Concentration (Cmax) for Ubrogepant Alone in Combination With Erenumab
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Ubrogepant Alone | Part 1: Ubrogepant in Combination With Erenumab
Number analyzed (Participants) | 20 | 19
ng/mL | 459.32 (168.56) | 486.80 (201.52)
Statistical Analysis 1: Comparison: Part 1: Ubrogepant Alone vs Part 1: Ubrogepant in Combination With Erenumab; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Mean Percentage = 103.86, 90% CI 2-sided [93.01 to 115.98] — Ratio of Geometric Mean Percentage=Ubrogepant in Combination with Erenumab/Ubrogepant Alone * 100

6. Primary Outcome: Part 2: Cmax for Ubrogepant Alone and in Combination With Galcanezumab
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2: Ubrogepant Alone | Part 2: Ubrogepant in Combination With Galcanezumab
Number analyzed (Participants) | 20 | 19
ng/mL | 415.34 (225.64) | 375.12 (152.08)
Statistical Analysis 1: Comparison: Part 2: Ubrogepant Alone vs Part 2: Ubrogepant in Combination With Galcanezumab; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of Geometric Mean Percentage = 99.55, 90% CI 2-sided [82.27 to 120.45] — Ratio of Geometric Mean Percentage=Ubrogepant in Combination with Galcanezumab/Ubrogepant Alone * 100

7. Secondary Outcome: Part 1: Time of Maximum Plasma Drug Concentration (Tmax) for Ubrogepant Alone and in Combination With Erenumab
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: Ubrogepant Alone | Part 1: Ubrogepant in Combination With Erenumab
Number analyzed (Participants) | 20 | 19
hour | 1.50 [1.00 to 3.00] | 1.48 [0.50 to 3.02]

8. Secondary Outcome: Part 2: Tmax for Ubrogepant Alone and in Combination With Galcanezumab
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Part 2: Ubrogepant Alone | Part 2: Ubrogepant in Combination With Galcanezumab
Number analyzed (Participants) | 20 | 19
hour | 1.50 [1.00 to 6.00] | 1.50 [0.98 to 6.00]

9. Secondary Outcome: Part 1: Terminal Elimination Rate Constant (λz) for Ubrogepant Alone and in Combination With Erenumab
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Part 1: Ubrogepant Alone | Part 1: Ubrogepant in Combination With Erenumab
Number analyzed (Participants) | 20 | 19
1/hour | 0.136 (0.025) | 0.156 (0.034)

10. Secondary Outcome: Part 2: λz for Ubrogepant Alone and in Combination With Galcanezumab
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/hour
Groups:
- Part 2: Ubrogepant Alone: Participant received Intervention A (ubrogepant 100 mg tablet) orally once daily on Day 1 under fasting conditions.
Arm/Group | Part 2: Ubrogepant Alone | Part 2: Ubrogepant in Combination With Galcanezumab
Number analyzed (Participants) | 20 | 19
1/hour | 0.150 (0.053) | 0.165 (0.056)

11. Secondary Outcome: Part 1: Terminal Elimination Half-life (T½) for Ubrogepant Alone and in Combination With Erenumab
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part 1: Ubrogepant Alone | Part 1: Ubrogepant in Combination With Erenumab
Number analyzed (Participants) | 20 | 19
hour | 5.26 (1.00) | 4.62 (0.94)

12. Secondary Outcome: Part 2: T½ for Ubrogepant Alone and in Combination With Galcanezumab
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part 2: Ubrogepant Alone | Part 2: Ubrogepant in Combination With Galcanezumab
Number analyzed (Participants) | 20 | 19
hour | 5.04 (1.47) | 4.60 (1.35)

13. Secondary Outcome: Part 1: Apparent Total Body Clearance of Drug From Plasma After Extravascular Administration (CL/F) for Ubrogepant Alone and in Combination With Erenumab
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | Part 1: Ubrogepant Alone | Part 1: Ubrogepant in Combination With Erenumab
Number analyzed (Participants) | 20 | 19
liter/hour | 57.35 (17.20) | 54.74 (16.27)

14. Secondary Outcome: Part 2: CL/F for Ubrogepant Alone and in Combination With Galcanezumab
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | Part 2: Ubrogepant Alone | Part 2: Ubrogepant in Combination With Galcanezumab
Number analyzed (Participants) | 20 | 19
liter/hour | 72.90 (38.07) | 68.94 (28.12)

15. Secondary Outcome: Part 1: Apparent Volume of Distribution During the Terminal Phase After Extravascular Administration (Vz/F) for Ubrogepant Alone in Combination With Erenumab
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Part 1: Ubrogepant Alone | Part 1: Ubrogepant in Combination With Erenumab
Number analyzed (Participants) | 20 | 19
liter | 436.95 (158.11) | 375.84 (161.42)

16. Secondary Outcome: Part 2: Vz/F for Ubrogepant Alone in Combination With Galcanezumab
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Part 2: Ubrogepant Alone | Part 2: Ubrogepant in Combination With Galcanezumab
Number analyzed (Participants) | 20 | 19
liter | 568.66 (497.92) | 449.26 (213.84)

17. Secondary Outcome: Number of Participants Who Had Potentially Clinically Significant (PCS) Postbaseline Vital Sign Values
Description: Vital Signs included assessments of Blood Pressure, Pulse Rate, Weight, Respiratory Rate and Temperature. The investigator determined if the postbaseline Vital Sign values were potentially clinically significant using the Vital Sign PCS Criteria in the Statistical Analysis Plan (SAP).
Time Frame: End of Dosing (EOD): Within 7 days of Day 16 or at the time of early termination (Up to Day 16)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (Intervention A Then B Then D) | Part 2 (Intervention A Then C Then D)
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

18. Secondary Outcome: Number of Participants Who Had PCS Postbaseline Laboratory Values
Description: Laboratory assessments included Chemistry, Hematology and Urinalysis tests. The investigator determined if the postbaseline laboratory results were potentially clinically significant using the Clinical Laboratory PCS Criteria in the SAP. Assessments of Chemistry only were collected at the Final Follow-up Visit
Time Frame: EOD: Within 7 days of Day 16 or at the time of early termination (Up to Day 16); Follow-up Visit 30 days after last dose (Up to Day 45 +/-3 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (Intervention A Then B Then D) | Part 2 (Intervention A Then C Then D)
Number analyzed (Participants) | 20 | 20
Participants
  Hematology; EOD | 0 | 1
  Chemistry; EOD | 0 | 0
  Chemistry; Follow-up Visit | 1 | 1
  Urinalysis; EOD | 1 | 0

19. Secondary Outcome: Number of Participants Who Had PCS Postbaseline Physical Examination Values
Time Frame: EOD: Within 7 days of Day 16 or at the time of early termination (Up to Day 16)
Population: As per the SAP, abnormalities in physical examinations during the study were captured in medical history or Adverse Events (AEs) data panels. Therefore, there were no separate analyses for physical examination planned.
Arm/Group | Part 1 (Intervention A Then B Then D) | Part 2 (Intervention A Then C Then D)
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Number of Participants Who Had PCS Postbaseline Electrocardiogram (ECG) Values
Description: A standard 12-lead ECG was performed. The investigator determined if the ECG postbaseline values were potentially clinically significant using the ECG PCS Criteria in the SAP.
Time Frame: EOD: Within 7 days of Day 16 or at the time of early termination (Up to Day 16)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (Intervention A Then B Then D) | Part 2 (Intervention A Then C Then D)
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

21. Secondary Outcome: Number of Participants With Adverse Events (AEs) by Severity, Related AEs and AEs Leading to Discontinuation
Description: An AE is any untoward medical occurrence in a patient or a participant using an investigational drug, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. The investigator determined if the AE was causally related to treatment. The investigator determined if the severity of the AE was Mild (transient with minimal intervention that does not interfere with usual activities), Moderate ( usually alleviated with an intervention, interferes with usual activities causing discomfort but does not cause permanent harm) or Severe (interrupts usual activities, affects clinical status or requires intensive intervention).
Time Frame: First dose to within 30 days after last dose (Up to Day 45 +/-3 days)
Population: Safety population included all participants who received/took at least 1 administration of study intervention. Data is reported by intervention actually received.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Intervention A (Ubrogepant): Intervention A (ubrogepant 100 mg tablet) single oral dose on Day 1 under fasted conditions.
- Part 1: Intervention B (Erenumab): Intervention B (erenumab 140 mg) single SC injection on Day 8.
- Part 1: Intervention D (Ubrogepant); Part 2: Intervention D (Ubrogepant): Intervention D (ubrogepant 100 mg tablet) orally once daily on Days 12, 13, 14 and 15 under fasted conditions.
- Part 2: Intervention A (Ubrogepant): Intervention A (ubrogepant 100 mg tablet) orally once daily on Day 1 under fasted conditions.
- Part 2: Intervention C (Galcanezumab): Intervention C (galcanezumab 120 mg) two SC injections on Day 8.
Arm/Group | Part 1: Intervention A (Ubrogepant) | Part 1: Intervention B (Erenumab) | Part 1: Intervention D (Ubrogepant) | Part 2: Intervention A (Ubrogepant) | Part 2: Intervention C (Galcanezumab) | Part 2: Intervention D (Ubrogepant)
Number analyzed (Participants) | 20 | 19 | 19 | 20 | 20 | 19
Participants
  All AEs | 7 | 8 | 7 | 2 | 3 | 4
  AEs by Severity: Mild | 7 | 8 | 6 | 2 | 3 | 4
  AEs by Severity: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  AEs by Severity: Severe | 0 | 0 | 1 | 0 | 0 | 0
  Related AEs | 2 | 7 | 5 | 0 | 3 | 3
  AEs Leading to Discontinuation | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose to within 30 days after last dose (Up to Day 45 +/-3 days)
Description: Safety population included all participants who received/took at least 1 administration of study intervention. Data is presented by intervention actually received.
Groups:
- Part 2; Intervention A (Ubrogepant): Intervention A (ubrogepant 100 mg tablet) orally once daily on Day 1 under fasted conditions.
Arm/Group | Part 1: Intervention A (Ubrogepant) | Part 1: Intervention B (Erenumab) | Part 1: Intervention D (Ubrogepant) | Part 2; Intervention A (Ubrogepant) | Part 2: Intervention C (Galcanezumab) | Part 2: Intervention D (Ubrogepant)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/19 | 0/20 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/19 | 0/20 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 7/20 | 8/19 | 7/19 | 2/20 | 3/20 | 4/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Intervention A (Ubrogepant) (N=20) | Part 1: Intervention B (Erenumab) (N=19) | Part 1: Intervention D (Ubrogepant) (N=19) | Part 2; Intervention A (Ubrogepant) (N=20) | Part 2: Intervention C (Galcanezumab) (N=20) | Part 2: Intervention D (Ubrogepant) (N=19)
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Puncture site pain (General disorders) | 3 | 0 | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 6 | 1 | 0 | 3 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT04179474/SAP_000.pdf
  • Study Protocol (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT04179474/Prot_001.pdf